CLINICAL TRIAL: NCT06645717
Title: Neuromotor Development in Children Enrolled in the Swedish Neonatal Follow-up Program and Access to Motor Related Healthcare
Brief Title: Neuromotor Development and Motor Related Health Care in Children with a High Risk Neonatal Period
Status: Not yet recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Maria Örtqvist, Associate professor, physiotherapist, Karolinska Institutet
Other Study IDs: 2024-01633-01
Record Dates: First submitted 2024-10-01; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Motor Disorders; Neurodevelopmental Disorders; Premature Birth; Hypoxic-Ischemic Encephalopathy; Small for Gestational Age At Delivery
Keywords: brain; HIE; SGA; preterm; neurodevelopment; motor related healthcare; children; motor function
MeSH Terms: conditions — Motor Disorders; Neurodevelopmental Disorders; Premature Birth; Hypoxia-Ischemia, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The overall aim of the study is to evaluate the prevalence of motor- and neurological disorders (cerebral pares and other less severe motor disorders) in Swedish infants with a high-risk neonatal period and to elucidate whether these children receive motor related health care (MRHC) at 2 and or 5,5 years of age.

DETAILED DESCRIPTION:
Specific aims:

1. To evaluate the prevalence of cerebral pares (CP) and other motor impairments in Swedish infants with a high-risk neonatal period (total group and sub-groups), followed up at age 2 and or 5,5 years.
2. To study how retinopathy of prematurity (ROP) affects the risk for later gross and fine motor impairments in children with a high-risk neonatal period, with specific reference to children born extremely preterm.
3. To study the number of children, with a high-risk neonatal period having access to MRHC (defined as having at least one visit over the previous year to a physiotherapist and/or an occupational therapist).

   * To evaluate possible associations between receiving MRHC and maternal-, pregnancy- and neonatal factors.
   * To study the association between receiving MRHC and cognition, motor function, behavior, quality of life and autism spectrum disorders (ASD) at age 2 and 5,5 years.
4. To study if there are regional differences in Sweden in follow-up of CP and less severe motor disorders at the age of 2 and 5,5 years.
5. To assess the completeness and agreement of some developmental and motor disorders, neurosensory impairments and chronical diseases in the Swedish Neonatal Quality Register (SNQ) with the Swedish National Patient Register (NPR) and The Cerebral Palsy Follow-Up Program (CPUP).

ELIGIBILITY:
Inclusion Criteria:

* Included in the SNQ registry and having a follow-up protocol for 2 and/or 5 years of age.

Exclusion Criteria:

* None if the above inclusion criteria ar true.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Today, data from 2,900 children are available in the follow-up protocol for 5,5 years of age in the SNQ according to the vice registry manager for the SNQ registry (Stellan Håkansson 08-03-2023).
Sampling Method: Non-Probability Sample
Enrollment: 2900 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2034-10-01 (Estimated)

PRIMARY OUTCOMES:
Movement assessment battery for children Second Edition (MABC-2) | Until 2026-10-01
  The MABC-2 is designed to identify and describe motor disorders in children and adolescents, from three to sixteen years of age. It gives information about both gross and fine motor functioning. It consists of eight tasks/items that are aggregated into three components: (1) Manual dexterity, that tests fine motor skills through three tasks, (2) Aiming and catching evaluates aiming and catching skills through two tasks/items, (3) Balance assesses gross motor skills through three tasks.
  The scoring procedure includes transforming raw scores into age adjusted scaled scores (mean 10; SD 3) for each item. The scaled scores of items within the same component are summed to obtain a total component score which is then converted into a scaled score and a percentil rank. The scaled scores of alla items are then summed to provide a total motor score that is converted into a total scaled score and percentile. Higher scores indicate better performance.
Bayley Scales of Infant Development Third Edition (Bayley III) | Until 2026-10-01
  The Bayley-III is an assessment tool to identify developmental impairments from birth to the age of 3. It includes cognitive, language, motor (gross and fine), social-emotional and adaptive behavior scales. It is often used in research and clinical work. Raw scores of successfully completed items are converted to scale scores and to composite scores. These scores are used to determine the child's performance compared with norms taken from typically developing children of their age (in months).
Wechsler Preschool and Primary Scale of Intelligence Fourth Edition (WPPSI-IV) | Until 2026-10-01
  The WPPSI-IV is a measure of general cognitive development for preschoolers and young children. The test is divided in two age intervals, 2 years and 6 months to 3 years and 11 months, and from 4 years to 7 years and 7 months. The younger age interval is divided into three primary index scales, verbal comprehension index (VCI), visual spatial index (VSI), and working memory index (WMI) and the older age interval consists of five primary index scales VCI, VSI, WMI, fluid reasoning index (FRI), and processing speed index (PSI). These primary index scales put together give a full-scale intelligence quotient (FSIQ) score.
The developmental coordination disorder questionnaire 2007 (DCDQ'07) | Until 2026-10-01
  DCDQ-07 is a brief parent questionnaire designed to screen for coordination disorders in children between 5 and 15. The DCDQ-07 is considered a valid clinical screening tool for children who have coordination disorders. DCDQ-07 has been validated against MABC-2. The questionnaire consists of 15 questions with answers from 1-5. All the answers are summed up together to a total score in the end. The higher the total score the less likely the child has developmental coordination disorder.
Movement Assessment battery for children Secondary Edition (MABC-2 checklist) | Until 2026-10-01
  Parent and teacher reported MABC-2 checklist is a screening tool for motor impairments in children between 3 and 16 years of age. It meets standards for reliability and validity when used in research and every day clinical work.
  The checklist contains two 15-item sections. Section A evaluates movement in both a static and/or predictable environment. Section B evaluates movement in a dynamic and/or unpredictable environment. The items in both sections are rated on a four-point liket rating scale ranging from very well to not close. The MABC-2 checklist total motor score is the sum of the scores for the two sections; the higher the score; the poorer the performance.
Kidsscreen 10 | Until 2026-10-01
  Kidsscreen 10 is used to assess self-reported subjective health and the mental, psychological and social well-being of children between 7 to 17 years of age. The instrument has shown adequate psychometrics. Kidsscreen 10 provides a global health related quality of life (HRQoL) and is recommended for use in larger studies.
  The kid screen-10 score contains 10 items. Each item is answered on a 5-point response scale. The responses are coded so that higher indicate better HRQoL.
Pediatric Quality of Life Inventory - Family Impact Module (PedsQL) | Until 2026-10-01
  Pedsql - Family Impact Module was designed to measure the impact of pediatric chronic health on the family and parents. This module encompasses six scales measuring parent self-reported functioning including physical, emotional, social and cognitive functioning, communication and worry. The module aslo measures parent-reported daily activities and family relationships. A 5-point response scale is used so that higher scores indicate better functioning.
MRHC motor related healthcare | Until 2026-10-01
  Receiving MRHC will be defined as having at least one visit to a physiotherapist and/or an occupational therapist during the previous year.
Study specific questionaire | Until 2026-10-01
  Study specific questionnaire about motor related health care and motor function. It consists of 6 main questions. The questionnaire does not give a total score but gives specific information about motor functioning, physical activity and visits to physiotherapists/pediatric neurologist/occupational therapist.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Örtqvist, PhD, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No